CLINICAL TRIAL: NCT07032844
Title: Comparing the Effectiveness of Primary Care Delivered Telehealth Interventions to Manage Type 2 Diabetes in People With Physical Disabilities and Multiple Chronic Conditions
Brief Title: Comparing Effectiveness of Primary Care-Delivered Telehealth Interventions to Manage Type 2 Diabetes in People With Physical Disabilities and Multiple Chronic Conditions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014522; TE-2023C3-34949 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-06-07; First posted 2025-06-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the study will receive one of the core interventions:
  1. Digital Health coaching
  2. Remote Patient Monitoring
  3. Combination of Digital Health coaching + Remote Patient Monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Health Coaching (Experimental): weekly coaching calls that address topics related to goal setting, creating supportive environments for behavior change, physical activity, and nutrition
  Interventions: Behavioral: Digital Health Coaching
- Remote Patient Monitoring (Experimental): Care coordinators within the RPM program will make individual contact with participants to discuss their plan and further educate on methods to manage their diabetes more efficiently.
  Interventions: Behavioral: Phone Based Coaching
- Combination of Digital Health Coaching and Remote Patient Monitoring (Experimental): Combination of Digital Health Coaching and Remote Patient Monitoring
  Interventions: Behavioral: Combination of Digital Health coaching + Remote Patient Monitoring

INTERVENTIONS:
Behavioral: Digital Health Coaching — This program will be developed using existing, evidence-based curricula for chronic disease self-management, with emphasis on diabetes, hypertension, and obesity. Prior to initiating health coaching with participants, coaches will review data collected related to SDoH to further tailor the intervention as appropriate for housing stability, access to food and transportation, and interpersonal safety. All coaches will have access to participants' EMRs such that they can view medical information throughout the intervention. Coaches will be trained using a curriculum developed by Family and Community Medicine's inter-professional care team and our partners at NCHPAD, making the coaching inclusive of people with physical disabilities, such that the coaches are proficient in motivating behavior change related to resilience, physical activity, nutrition, mindfulness, and relationship-building, among others.
  Arms: Digital Health Coaching
Behavioral: Phone Based Coaching — Weekly coaching calls that address topics related to goal setting, creating supportive environments for behavior change, physical activity, and nutrition.
  Arms: Remote Patient Monitoring
Behavioral: Combination of Digital Health coaching + Remote Patient Monitoring — Combination of both digital health coaching and remote patient monitoring
  Arms: Combination of Digital Health Coaching and Remote Patient Monitoring

SUMMARY:
The purpose of the study is to compare 2 primary care based telehealth interventions- 1) digital health coaching and 2) remote patient monitoring for improving glycemic (blood sugar levels) control and overall health outcomes in individuals with physical disabilities, type 2 diabetes (T2DM) and at least one chronic condition. The project aims to determine which intervention is more effective in reducing blood sugar levels, improving patient-reported outcomes such as diabetes-related distress, and facilitating the implementation of these approaches in real-world primary care settings serving vulnerable populations. The findings intend to inform about optimal telehealth strategies for managing multiple chronic conditions in underserved groups, there by supporting improved health equity and quality of care.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) defines chronic diseases as conditions that last one year or more and require ongoing medical attention, limit activities of daily living, or both. Six in 10 adults in the U.S. are reported to have at least one chronic condition, while four in 10 adults in the U.S. are reported to have two or more chronic conditions.T2DM is one of the chronic conditions in the U.S. population that has been gradually increasing over the years. Over 34.2 million U.S. adults are affected by diabetes mellitus (DM); T2DM accounts for 90-95% of these.T2DM is often associated with other cardiometabolic diseases such as hypertension and obesity.T2DM is one of the strongest risk factors for cardiovascular disease (CVD) and chronic kidney disease (CKD), which are among the leading causes of death in the U.S. T2DM also results in physical disability because of complications such as leg amputation and vision loss.

Individuals with physical disabilities face a disproportionate burden of T2DM and related chronic conditions, exacerbated by suboptimal social determinants of health (SDoH) such as reduced healthcare access and economic inequities.In general, 50-60% of disparities in T2DM outcomes can be attributed to social determinants of health (SDoH). SDoH are defined as the conditions in which people are born, grow, live, work, and age. Physical disability has an intimate relationship with SDoH such as race/ethnicity, sex, socioeconomic status, geographic location, access to and quality of healthcare, etc. Transformation from the status of able-bodied person to the status of disability leads to a disparity and decline in SDoH of these individuals in terms of geographic location, healthcare access, transportation, economic support, food security, and so on.

Teleheath interventions, including digital health coaching (DHC) and remote patient monitoring(RPM), have emerged as promising strategies to address these disaprtiites, improve glycemic control, and overcome barriers to care. Developing an optimal, interdisciplinary primary care delivery model incorporating digital health coaching or RPM may play a crucial role in overcoming the obstacle of suboptimal patient-physician communication by enhancing both physician and patient satisfaction and improving population health. Both digital health coaching and RPM address SDoH, are being implemented by health systems, and show evidence of effectiveness through trials as well as real-world effectiveness.

However, there exists a clear evidence gap about which of these two interventions are superior and will best optimize population health outcomes. Further, there is an evidence gap about how these telehealth interventions may help people with physical disabilities and multiple chronic conditions and affect their long-term outcomes. The project design addresses this critical gaps identified in earlier research. While both interventions (RPM and DHC) show promise individually, no direct comparisons exist in populations with physical disabilities- a group disproportionally affteced by diabtese and access barriers. Previous studies often excluded this demographic or focused on single chronic conditions, despite evidence that multimorbidity complicates self-management. Aditionally, implementation science gaps presists regarding workflow integration in real-world primary car settings serving vulnerable groups.

ELIGIBILITY:
Inclusion Criteria:

1. Physical Disability
2. Diagnosed with Type 2 Diabetes
3. Hemoglobin A1c ≥7% within 3 months of screening
4. Must have at least 1 additional chronic conditions from the list below Hypertension Congestive Heart Failure Coronary Artery Disease Hyperlipidemia Stroke Arthritis Asthma Cancer Chronic Kidney Disease (Stages 1-4) COPD Osteoporosis Multiple Sclerosis Parkinsons

Exclusion Criteria:

1. Intellectual, Learning, Developmental Disabilities
2. Non-english speakers
3. Currently pregnant
4. Significant vision loss preventing use of phone/tablet for interventions
5. Received Remote Patient Monitoring or Digital Health Coaching for T2DM management within 30 days of enrollment
6. End-stage kidney disease (on dialysis)
7. Does not report having a physical disability
8. Perceived unwillingness or inability to participate

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 12 months
  Our primary aim 1 compares the average treatment effectiveness of a six-month RPM, digital health coaching, and combination digital health coaching and RPM program through a multi-site pragmatic randomized trial design. Our primary outcome is reduction in HbA1c at 12 months. Investigators hypothesize that the combination arm will result in superior improvements in HbA1c compared to either intervention alone, aligning with preliminary stakeholder engagement suggesting patient-centered preference for this combined approach.

SECONDARY OUTCOMES:
Diabetes Distress Screening Scale Results | 12 months
  Investigators hypothesize that the combination arm will result in more significant improvements in diabetes distress compared to either the remote patient monitoring (RPM) or digital health coaching alone.

OTHER OUTCOMES:
Understand for Whom each intervention is more effective | 12 months
  To conduct pre-specified and exploratory predictive modeling that explains the heterogeneity in treatment effects and helps us understand for whom either of these interventions is more effective.
Identify the contextual factors that affect implementation of the different intervention components. | 12 months
  A convergent, mixed methods approach rooted in the Consolidated Framework for Implementation Research (CFIR) will be used to assess the multifaceted, multilevel relationships among context, intervention implementation processes, and implementation outcomes. Implementation outcomes of the intervention will be evaluated by the reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) framework.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Mehta, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided